CLINICAL TRIAL: NCT06100939
Title: A Multicenter, Randomized, Double-Masked, Sham-Controlled, Parallel-Group Phase 3 Study to Evaluate the Efficacy and Safety of Epithelium-On Corneal Cross-linking in Subjects 8 to 45 Years of Age With Keratoconus (APRICITY-A)
Brief Title: Epithelium-On Corneal Cross-linking in Subjects 8 to 45 Years of Age With Keratoconus
Acronym: Apricity-A
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Epion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CXL-006-A
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus | interventions — Riboflavin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active Treatment (Experimental): Epithelium-on corneal cross-linking
  Interventions: Combination Product: Riboflavin and Sodium Iodide solution and Ultraviolet-A treatment
- Control Treatment (Placebo Comparator): Placebo and sham for epithelium-on corneal cross-linking
  Interventions: Combination Product: Placebo and sham treatment

INTERVENTIONS:
Combination Product: Riboflavin and Sodium Iodide solution and Ultraviolet-A treatment — Drug: Ribostat riboflavin and sodium iodide ophthalmic solution
  Device: UV-3000 ultraviolet A light source
  Arms: Active Treatment
Combination Product: Placebo and sham treatment — Drug: placebo ophthalmic solution
  Device: UV-3000 light source
  Arms: Control Treatment

SUMMARY:
A Multicenter, Randomized, Double-Masked, Sham-Controlled, Parallel-Group Phase 3 Study to Evaluate the Efficacy and Safety of Epithelium-On Corneal Cross-linking in Subjects 8 to 45 Years of Age With Keratoconus

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of keratoconus

Exclusion Criteria:

* Minimal corneal thickness < 350 microns
* Non-keratoconic ectatic disease
* Contraindications or hypersensitivities to any required study medications
* Pregnancy or breastfeeding
* Certain concomitant ocular conditions

Ages: 8 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Best Spectacle-Corrected Distance Visual Acuity (BSCDVA) | Baseline to 12 months
  BSCDVA will be assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts. The score ranges from 0 to 100, with a higher score representing better visual functioning.

SECONDARY OUTCOMES:
Vision-related Quality of Life as Assessed by the National Eye Institute 25-Item Visual Function Questionnaire (NEI-VFQ-25) | Baseline to 12 months
  The score on the NEI-VFQ-25 ranges from 0 to 100, with a higher score indicating greater functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Belin, MD, Study Director — Epion Therapeutics
Locations (13):
- United States (13):
  - Nvision Eye Centers Rowland Heights, Rowland Heights, California
  - Goodman Eye Center, San Francisco, California
  - Center for Excellence in Eye Care, Miami, Florida
  - Chicago Cornea Consultants, Hoffman Estates, Illinois
  - Boston Vision, Brookline, Massachusetts
  - Ophthalmology Associates, St Louis, Missouri
  - The Eye Doctors at CNY Eye Care, East Syracuse, New York
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Devers Eye Institute, Portland, Oregon
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - UPMC Vision Institute, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No